CLINICAL TRIAL: NCT07285564
Title: Performance of 18F-FDG Micro-PET-CT in the Assessment of Surgical Margins in Head and Neck Cancer
Acronym: TEP Margins
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB25.06
Record Dates: First submitted 2025-11-21; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Head & Neck Cancer
Keywords: Margins; microPET/CT; specimen
MeSH Terms: conditions — Head and Neck Neoplasms; Margins of Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): PET/CT of the specimen after surgery
  Interventions: Device: micro PET/CT

INTERVENTIONS:
Device: micro PET/CT — PET/T of the speciment after surgery

SUMMARY:
The purpose of this study is to evaluate the diagnostic performance of 18F-FDG micro-PET-CT in malignant Head and neck cancer compared to definitive histological analysis (gold standard).

DETAILED DESCRIPTION:
In approximately 20% of cases, surgical margins are considered insufficient. The only tool currently available intraoperatively to assess the quality of surgical resection is the extemporaneous examination. This has a sensitivity of only 10%.

The objective is therefore to evaluate the performance of another tool, available intraoperatively, to help surgeons assess the quality of their resection. Currently, micro-PET-CT allows for the evaluation of surgical specimens (CE marking and FDA approval obtained). Its performance in the evaluation of surgical margins remains to be demonstrated. This is the subject of the present study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Adult, male or female, aged 18 or over
* Patient with a malignant tumor of the oral cavity, oropharynx, hypopharynx, larynx, sinuses, or salivary glands, regardless of lymph node status (any N) M0, operable
* Member or beneficiary of a social security plan

Exclusion Criteria:

* Child-Pugh C liver failure
* Patients under guardianship, conservatorship, or legal protection
* Patients deprived of their liberty
* Pregnant or breastfeeding women
* Hypersensitivity to 18F-FDG or any of its excipients (ethanol or water for injection)
* Uncontrolled diabetes
* Moderate to end-stage renal failure, stage IIIB to V (glomerular filtration rate less than 44 mL/min/1.73 m²)
* Patients unable to understand the study for any reason or to comply with the trial requirements (language, psychological, or geographical issues).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate the diagnostic performance of 18F-FDG micro-PET-CT in malignant ENT tumors compared to definitive histological analysis (gold standard). | Surgery
  Estimate the performance of micro-FDG PET in defining surgical margins and compare with histology by measuring the number of quadrants affected by each technique on the surgical specimen

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Hapdey, PhD, Principal Investigator — Centre Henri Becquerel; Lise-Marie Roussel, MD, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France